CLINICAL TRIAL: NCT01124695
Title: A Phase II Prospective Trial Correlating Progression Free Survival With CYP2D6 Activity in Patients With Metastatic Breast Cancer Treated With Single Agent Tamoxifen
Brief Title: Tamoxifen Citrate in Treating Patients With Metastatic or Recurrent Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E3108; E3108 (Other: ECOG-ACRIN Cancer Research Group); U10CA180794 (NIH)
Record Dates: First submitted 2010-05-14; First posted 2010-05-17 (Estimated); Results first posted 2023-03-14 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Stage IV Breast Cancer
Keywords: estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer; recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tamoxifen (Experimental): Patients receive oral tamoxifen citrate once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicities.
  Interventions: Drug: tamoxifen

INTERVENTIONS:
Drug: tamoxifen — PO
  Other Names: tamoxifen citrate; Nolvadex; NSC# 180973

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using tamoxifen citrate may fight cancer by blocking the use of estrogen by tumor cells.

PURPOSE: This phase II trial is studying how well tamoxifen citrate works in patients with metastatic or recurrent breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To correlate CYP2D6 (Cytochrome P450 2D6) score (0 vs 1-2) and progression-free survival (PFS)

Secondary

* To correlate CYP2D6 score (0 vs 1 vs 2) and PFS
* To correlate CYP2D6 score (0 vs 1-2) and the proportion of these patients who are progression-free at 6 months.
* To correlate endoxifen concentration with response
* To correlate CYP2D6 with response
* To correlate the presence of candidate estrogen receptor (ESR) 1 and 2 variant alleles, UDP-glucuronosyltransferases (UGT) 7, sulfotransferases (SULT) 1A1, other candidate genes and biomarkers to PFS and other tamoxifen related outcomes

OUTLINE: This is a multicenter study.

Patients receive oral tamoxifen citrate once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicities.

Blood, plasma, and tissue samples are collected periodically for laboratory studies.

After completion of study therapy, patients are followed up every 3-6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the breast

  * Stage III (locally advanced), metastatic, or recurrent disease
  * Deemed not resectable
* Estrogen-receptor and/or progesterone-receptor positive disease

  * Receptor status is based on most recent results
* Measurable or non-measurable disease
* ECOG performance status 0-2
* History of central nervous system (CNS) metastasis allowed provided it has been treated (surgery, radiotherapy, or radiosurgery) within the past 4 weeks and does not require medications to control symptoms
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 times ULN (≤ 5 times ULN if liver metastases present)
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception
* Disease-free of prior invasive malignancies for ≥ 5 years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Prior chemotherapy, trastuzumab, or bevacizumab in the adjuvant setting allowed provided it has been completed ≥ 4 weeks before study therapy; other prior non-hormonal investigational agents in the adjuvant setting must have been completed at least 4 weeks prior to study registration and should be discussed with the study PI
* Prior tamoxifen as adjuvant treatment is allowed as long as the patient did not have disease relapse or progression while on adjuvant tamoxifen or within 4 weeks of last dose
* Treatment in the advanced setting must have been completed at least 2 weeks prior to study initiation
* Prior aromatase inhibitors (e.g., anastrozole, letrozole, exemestane, aminoglutethamide) are allowed in the adjuvant or metastatic setting
* At least 2 weeks since prior and no concurrent medications that are strong to moderate inhibitors of CYP2D6 and may alter tamoxifen citrate metabolism including, but not limited to, any of the following:

  * Paroxetine (Paxil)
  * Fluoxetine (Prozac)
  * Bupropion (Wellbutrin)
  * Quinidine (Cardioquin)
* Concurrent radiotherapy to painful sites of bone disease or areas of impending fractures allowed provided the following criteria are met:

  * Radiotherapy was initiated before study entry
  * Sites of measurable or non-measurable disease are outside the radiotherapy port
  * Recovered from prior radiotherapy

Exclusion Criteria:

* Pregnant or nursing
* Concurrent chemotherapy
* Leptomeningeal disease
* Non-protocol concurrent hormonal therapy
* Medical or psychiatric conditions that would interfere with protocol compliance, the ability to provide informed consent, assessment of response, or anticipated toxicities
* Prior tamoxifen for advanced disease
* More than 2 lines of non-hormonal treatment in the locally advanced or metastatic setting, including trastuzumab (Herceptin), bevacizumab, or other biologics
* Starting bisphosphonate therapy while receiving treatment on this study

  * Patients who have begun receiving bisphosphonate therapy prior to registration may continue at the same intervals used prior to study registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-01-07 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (294):
- United States (292):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - Mercy Cancer Center at Mercy Medical Center, Merced, California
  - Camino Medical Group - Treatment Center, Mountain View, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - University of California Davis Cancer Center, Sacramento, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Central Care Cancer Center at Carrie J. Babb Cancer Center, Bolivar, Missouri
  - Skaggs Cancer Center at Skaggs Regional Medical Center, Branson, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Mercy Clinic Cancer and Hematology - Rolla, Rolla, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center - South, Las Cruces, New Mexico
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - St. Luke's - Roosevelt Hospital Center - St.Luke's Division, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Cleveland Clinic Beachwood Family Health and Surgery Center, Beachwood, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Cleveland Clinic Foundation - Strongsville, Strongsville, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Cancer Care Associates - Norman, Norman, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Doylestown Hospital Cancer Center, Doylestown, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Island Hospital Cancer Care Center at Island Hospital, Anacortes, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Highline Medical Center Cancer Center, Burien, Washington
  - Swedish Medical Center - Issaquah Campus, Issaquah, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic - Marinette, Marinette, Wisconsin
  - D.N. Greenwald Center, Mukwonago, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
- British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia, Canada
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Derived] Stearns V, ONeill A, Schneider BP, Skaar TC, Liu MC, Lohrisch C, Goetz MP, Vallejos CS, Sparano JA, Villa D, Silverman P, Cheema PS, Moore DF Jr, Sledge GW Jr. CYP2D6 activity in patients with metastatic breast cancer treated with single agent tamoxifen: results from ECOG-ACRIN E3108. Breast Cancer Res Treat. 2025 Feb;209(3):595-602. doi: 10.1007/s10549-024-07519-z. Epub 2024 Oct 21. PMID 39432161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on September 21, 2010, accrued its first patient on January 7, 2011, and closed on October 22, 2015 for a total of 124 patients enrolled.
Groups:
- Tamoxifen: Patients receive oral tamoxifen citrate at 20 mg once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicities.
Period: Overall Study
Arm/Group | Tamoxifen
Started | 124
Treated | 122
Eligible and Treated | 113
Eligible and Treated and Had CYP2D6 Score | 85
Eligible and Treated and Had Cycle 3 Edoxifen Evaluation | 63
Eligible and Treated Patients With 3-month Endoxifen and Were Progression-free and Alive at 3 Months | 43
Completed | 1
Not Completed | 123
Not completed — Disease progression | 77
Not completed — Adverse Event | 11
Not completed — Death | 1
Not completed — Withdrawal by Subject | 7
Not completed — Physician Decision | 3
Not completed — Alternative therapy | 9
Not completed — No documentation that patient went off treatment | 4
Not completed — Ineligible | 9
Not completed — Ineligible and never start treatment | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients are included in this analysis. This is the primary analysis population.
Arm/Group | Tamoxifen
Number analyzed (Participants) | 113
Age, Continuous [Median (Full Range); unit: years] | 62 [36 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33
  Not Hispanic or Latino | 77
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 97
  More than one race | 0
  Unknown or Not Reported | 3
CYP2D6 phenotype [Count of Participants; unit: Participants]
  Poor metabolizer | 2
  Intermediate metabolizer | 27
  Normal metabolizer | 50
  Ultra-rapid metabolizer | 6
  Missing | 28

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival by CYP2D6 Status in 2 Categories
Description: Progression-free survival is defined as the time from registration to progression or death, whichever occurs first. Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) was used to evaluate progression. Progression is defined as appearance of one or more new lesions or unequivocal progression of existing non-target lesions or at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Assessed every 3 months for 2 years, then every 6 months up to 5 years
Population: Eligible and treated patients who had a sample from baseline evaluable for CYP2D6 phenotype
Measure: Median (95% Confidence Interval); unit: months
Groups:
- CYP2D6 - PM: Patients with CYP2D6 score of 0 are considered as poor metabolizer (PM).
- CYP2D6 - (IM+NM+UM): Patients with CYP2D6 score >0 are included in the IM+NM+UM group.
  Intermediate metabolizer (IM): CYP2D6 score >0 and <=1 Normal metabolizer (NM): CYP2D6 score >1 and <=2 Ultra-rapid metabolizer (UM): CYP2D6 score >2
Arm/Group | CYP2D6 - PM | CYP2D6 - (IM+NM+UM)
Number analyzed (Participants) | 2 | 83
months | 12.9 [NA to NA] — Only 2 patients were in this category. Among these two, one was censored at baseline. As only one patient contributed data, the 95% CI could not be calculated. | 6.9 [4.4 to 8.5]

2. Secondary Outcome: Progression-free Survival by CYP2D6 Status in 3 Categories
Description: as for outcome 1
Time Frame: Assessed every 3 months for 2 years, then every 6 months up to 5 years
Population: Eligible and treated patients who had a sample from baseline evaluable for CYP2D6 phenotype
Measure: Median (95% Confidence Interval); unit: months
Groups:
- CYP2D6 - IM: Intermediate metabolizer (IM): CYP2D6 score >0 and <=1
- CYP2D6 - NM+UM: Patients with CYP2D6 score >1 are included in the NM+UM group.
  Normal metabolizer (NM): CYP2D6 score >1 and <=2 Ultra-rapid metabolizer (UM): CYP2D6 score >2
Arm/Group | CYP2D6 - PM | CYP2D6 - IM | CYP2D6 - NM+UM
Number analyzed (Participants) | 2 | 27 | 56
months | 12.9 [NA to NA] — Only 2 patients were in this category. Among these two, one was censored at baseline. As only one patient contributed data, the 95% CI could not be calculated. | 4.8 [2.7 to 13.8] | 7.4 [4.9 to 10.3]

3. Secondary Outcome: Proportion of Patients Progression-free at 6 Months
Description: Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) was used to evaluate progression. Progression is defined as appearance of one or more new lesions or unequivocal progression of existing non-target lesions or at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Assessed every 3 months for 6 months
Population: Eligible and treated patients who had a sample from baseline evaluable for CYP2D6 phenotype
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | CYP2D6 - PM | CYP2D6 - (IM+NM+UM)
Number analyzed (Participants) | 2 | 83
proportion of participants | 1.0 [0.16 to 1.00] | 0.50 [0.39 to 0.62]

4. Secondary Outcome: Proportion of Patients With Response
Description: Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) was used to evaluate response. Either complete response (CR) or partial response (PR) is considered as response. CR is defined as disappearance of all lesions. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Assessed every 3 months for 2 years, then every 6 months up to 5 years
Population: Eligible and treated patients who had a sample from baseline evaluable for CYP2D6 phenotype
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | CYP2D6 - PM | CYP2D6 - (IM+NM+UM)
Number analyzed (Participants) | 2 | 83
proportion of participants | 0 [0.0 to 0.84] | 0.13 [0.07 to 0.22]

5. Secondary Outcome: Endoxifen Concentration by Response
Description: Endoxifen (ng/ml) was assessed at cycle 3.
  Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) was used to evaluate response. Either complete response (CR) or partial response (PR) is considered as response. CR is defined as disappearance of all lesions. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Endoxifen was assessed at cycle 3; response was assessed every 3 months for 2 years, then every 6 months up to 5 years
Population: Eligible and treated patients who had a sample at cycle 3 for endoxifen concentration evaluation
Measure: Median (Full Range); unit: ng/ml
Groups:
- Responders: Patients with CR or PR per RECIST 1.1
- Non-responders: Patients without CR or PR per RECIST 1.1
Arm/Group | Responders | Non-responders
Number analyzed (Participants) | 6 | 57
ng/ml | 17.5 [7.5 to 45.2] | 17.2 [2.0 to 67.9]

6. Secondary Outcome: Progression-free Survival From 3 Months Post Registration
Description: This is a landmark progression-free survival analysis at 3 months post registration. Only patients who were progression-free and alive at 3 months were included.
  Progression-free survival in this analysis is defined as the time from 3 months post registration to progression or death, whichever occurs first. Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1) was used to evaluate progression. Progression is defined as appearance of one or more new lesions or unequivocal progression of existing non-target lesions or at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Assessed every 3 months for 2 years, then every 6 months up to 5 years
Population: Eligible and treated patients who had endoxifen level assessed at 3 months and were progression-free and alive at 3 months from registration
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Endoxifen High: Patients with endoxifen at 3 months higher than median (15.5 ng/ml)
- Endoxifen Low: Patients with endoxifen at 3 months lower than or equal to median (15.5 ng/ml)
Arm/Group | Endoxifen High | Endoxifen Low
Number analyzed (Participants) | 21 | 22
months | 13.8 [6.5 to 16.6] | 11.1 [5.3 to 19.3]

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment up to 5 years
Description: All patients enrolled are included in all-cause mortality analysis. Patients who received treatment with adverse event data available are included in AE analysis.
  This is a single-arm study, so adverse events are reported for the Tamoxifen arm only, which is reported per arm.
Arm/Group | Tamoxifen
All-Cause Mortality (participants affected / at risk) | 69/124
Serious Adverse Events (participants affected / at risk) | 30/122
Other Adverse Events (participants affected / at risk) | 18/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tamoxifen (N=122)
Anemia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 2
Aspartate aminotransferase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 2
Pericardial tamponade (Cardiac disorders) | 1
Death NOS (General disorders) | 1
Edema limbs (General disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Joint infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Weight gain (Investigations) | 1
White blood cell decreased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Neoplasms - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Confusion (Psychiatric disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Chronic kidney disease (Renal and urinary disorders) | 1
Surgical and medical procedures - Other (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tamoxifen (N=122)
Fatigue (General disorders) | 18
Hot flashes (Vascular disorders) | 11
Anemia (Blood and lymphatic system disorders) | 10
Edema limbs (General disorders) | 8
Constipation (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 9
Aspartate aminotransferase increased (Investigations) | 8
Anorexia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 17
Bone pain (Musculoskeletal and connective tissue disorders) | 8
Anxiety (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Hypertension (Vascular disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT01124695/Prot_SAP_000.pdf